CLINICAL TRIAL: NCT05979103
Title: Music Genre Stereotypes to Boost Relaxation in Chronic Pain Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Sean D Young, Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3585
Record Dates: First submitted 2023-07-28; First posted 2023-08-07 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Reggae Music (Experimental): Group 1 (Reggae): Participants in this group will be told about he stereotype of reggae in making people more calm. They will listen to reggae music over the 4 weeks.
  Interventions: Behavioral: Listening to Reggae Music and told the stereotype
- Preferred Music (Active Comparator): Group 2 (Preferred): Participants in this group will listen to preferred music over the 4 weeks and will not be told any stereotypes.
  Interventions: Behavioral: Listening to Preferred Music
- Control (No Intervention): Group 3 (Waitlist- Control): Participants are not providing with any intervention. They only complete surveys.

INTERVENTIONS:
Behavioral: Listening to Reggae Music and told the stereotype — Participants in this group will be told about he stereotype of reggae in making people more calm. They will listen to reggae music over the 4 weeks. Each day, we will send them a playlist to listen to.
  Arms: Reggae Music
Behavioral: Listening to Preferred Music — Participants in this group will NOT be told the stereotype for the audio they are listening to. They will listen to preferred music over the 4 weeks. Each day, we will remind them to listen to preferred music.
  Arms: Preferred Music

SUMMARY:
Social psychological research has demonstrated that internalized stereotypes affect people's attitudes and behaviors. Music-based interventions that rely on stereotypes might have promise for keeping participants engaged in health interventions, reducing stress, and improving wellbeing.

DETAILED DESCRIPTION:
Group Assignments

Participants will be randomized into one of four groups.

1. Group 1 (Reggae): Participants in this group will receive the stereotype and listen to the music over the 4 weeks.
2. Group 2 (Preferred): Participants in this group will listen to preferred music over the 4 weeks.
3. Control Group: Participants in this group will serve as a control and will not receive any intervention until the study is completed. They will complete a baseline survey and a follow-up survey at four weeks, as well as similar daily surveys. Some recordings will be sent to this group after the study is completed, without tracking their usage.

Intervention

All groups will complete a baseline and 4-week follow-up survey.

Participants in Group 1 and Group 2 will engage in daily listening 4-week intervention.They will have access to electronic audio recordings, with the order of listening labeled for each day. It is up to them if they want to listen to the daily recordings.

ELIGIBILITY:
Inclusion Criteria:

1. Are 18+
2. Live in the US
3. Are an English-proficient adult with a chronic pain diagnosis (no restrictions placed on type)
4. Have a pain rating of four or greater in average pain on a 0-10 numeric rating scale in the preceding week
5. Have had pain for at least 3 months and for at least 15 days in the preceding 30 days
6. Have moderate to severe anxiety based on GAD-7

Exclusion Criteria:

1. Are currently using or have used prescription opioids in the past 3 months to minimize a known treatment confound and increase sample homogeneity
2. Have a current cancer diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Generalized Anxiety Disorder (GAD-7) Score | 4 weeks
  Anxiety levels will be evaluated using the General Anxiety Disorder (GAD-7) questionnaire. Range 0-21, where higher score is greater anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California Irvine, Irvine, California, United States